CLINICAL TRIAL: NCT04885751
Title: Compare the Effect of Eupatilin and Rebamipide on the Prevention of Gastroenteropathy in Patients With NSAIDs and Low Dose Steroid: A Single-center, Randomized, Open Labeled, Pilot Study
Brief Title: Compare the Effect of Eupatilin and Rebamipide on the Prevention of Gastroenteropathy
Acronym: CEERS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Boramae Hospital (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hyoun Woo Kang, Associate professor, Seoul National University Boramae Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Eupatilin_GEP_01
Record Dates: First submitted 2021-04-26; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Ankylosing Spondylitis; Other Musculoskeletal Disorder; Gastric Ulcer; Enteritis; NSAID-Associated Gastropathy; NSAID (Non-Steroidal Anti-Inflammatory Drug) Induced Enteropathy
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Spondylitis, Ankylosing; Stomach Ulcer; Enteritis | interventions — eupatilin; rebamipide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eupatilin (Experimental): take eupatilin to prevent NSAID induced gastroenteropathy
  Interventions: Drug: Eupatilin
- rebamipide (Active Comparator): take rebamipide to prevent NSAID induced gastroenteropathy
  Interventions: Drug: Rebamipide

INTERVENTIONS:
Drug: Eupatilin — take eupatilin to prevent NSAID induced gastroenteropathy
  Arms: eupatilin
Drug: Rebamipide — take rebamipide to prevent NSAID induced gastroenteropathy
  Arms: rebamipide

SUMMARY:
The purpose of this study is to evaluate the efficacy of eupatilin on the prevention of gastroenteropathy in patients with NSAIDs and low dose steroid by comparing with rebamipide.

DETAILED DESCRIPTION:
After being informed of the study and potential risks, all patients giving written informed consents will undergo a 1-week screening period to determine eligibility for study entry. During screening period, patients will undergo fecal calprotectin test, upper endoscopy and submit symptom diary. At week 0, subjects who meet the eligibility criteria will be randomized in a open labeled manner in 1:1 ratio to eupatilin (90mg twice daily-test group, 25 patients) or rebamipide (100mg three times daily-control group paients) for 8 weeks. At week 8, subjects undergo fecal calprotectin test, upper endoscopy and submit symptom diary.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women who were adults at the time of receipt of written consent (age 19-70)
2. Those with rheumatoid arthritis, osteoarthritis, ankylosing spondylitis, or other musculoskeletal diseases that require continuous administration of nonsteroidal anti-inflammatory drugs (NSAIDs) and oral steroids for more than 8 weeks.
3. At screening (before baseline) endoscopy results Modified Lanza Score (MLS) 0~2
4. Those who have not had severe gastrointestinal symptoms in the previous 3 months[Excluding mild abdominal distention, abdominal pain, diarrhea, dyspepsia, nausea, and vomiting]
5. A person who agrees to participate in this clinical trial and voluntarily signs a written consent form

Exclusion Criteria:

1. Those with a history of gastrointestinal surgery (excluding appendectomy)
2. Those who have a history of esophageal cancer, liver cancer, pancreatic cancer, gastric cancer, colon cancer, small intestine tumor or other malignant disease within 5 years from the time of screening
3. Gastrointestinal diseases that are clinically significant by upper gastrointestinal endoscopy, namely active peptic ulcer, reflux esophagitis, gastroesophageal varices, Barrett's esophagus, Barrett's esophagitis, esophageal stenosis, inflammatory bowel disease (Those diagnosed with inflammatory bowel disease, IBD), gastrointestinal bleeding, etc.
4. Those with a history of recurrent gastrointestinal ulcer/perforation
5. Those with cerebrovascular bleeding or confirmed systemic bleeding disorder
6. Persons with severe uncontrolled heart failure (NYHA Class III-IV), high blood pressure (above 160/100 mmHg)
7. Those who have plans for surgical operation during the clinical trial period
8. Persons with a history of chronic pancreatitis, chronic renal diseases, chronic liver diseases, or other serious comorbid diseases
9. Those with clinically significant abnormal values (AST, ALT, BUN, Cr exceeding 2.5 times or Hb<10g/dL) by laboratory examination
10. Those with a history of alcohol or drug abuse/dependence
11. Pregnant and lactating women
12. Those who participated in other clinical trials within 30 days prior to participation in this clinical trial and received investigational drugs or received procedures
13. Patients who are difficult to perform this clinical trial by other investigators or who are judged to have medical findings that are not suitable for the clinical trial
14. Those who received celecoxib and prednisolone (or methylprednisolone) within 30 days prior to participation in this clinical trial

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with gastric damage | evaluated at day 56
  Percentage of patients with endoscopic Modified Lanza Score >3

SECONDARY OUTCOMES:
Change of gastric erosion number | evaluated at day 0 and day 56
  Change of gastric erosion number at day 56 compared with that at day 0
Change of Modified Lanza Score | evaluated at 0 day and day 56
  Change of Modified Lanza Score at day 56 compared with that at day 0
Change of duodenal erosion number | evaluated at day 0 and day 56
  Change of duodenal erosion number at day 56 compared with that at day 0
Gastrointestinal symptom | evaluated at day 0 and day 56
  Gastrointestinal symptom change using survey at day 56 compared with that at day 0
Fecal calprotectin | evaluated at day 0 and day 56
  Fecal calprotectin level change at visit 3 compared with visit 0
Antioxidant gene expression | evaluated at day 0 and day 56
  Antioxidant gene expression change at day 56 compared with that at day 0

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Sperling RL. NSAIDs. Home Healthc Nurse. 2001 Nov;19(11):687-9. doi: 10.1097/00004045-200111000-00011. No abstract available. PMID 12035587
- [Background] Conaghan PG. A turbulent decade for NSAIDs: update on current concepts of classification, epidemiology, comparative efficacy, and toxicity. Rheumatol Int. 2012 Jun;32(6):1491-502. doi: 10.1007/s00296-011-2263-6. Epub 2011 Dec 23. PMID 22193214
- [Background] MacDonald TM. Epidemiology and pharmacoeconomic implications of non-steroidal anti-inflammatory drug-associated gastrointestinal toxicity. Rheumatology (Oxford). 2000 Dec;39 Suppl 2:13-20; discussion 57-9. doi: 10.1093/rheumatology/39.suppl_2.13. PMID 11276797
- [Background] Lee SH, Han CD, Yang IH, Ha CW. Prescription pattern of NSAIDs and the prevalence of NSAID-induced gastrointestinal risk factors of orthopaedic patients in clinical practice in Korea. J Korean Med Sci. 2011 Apr;26(4):561-7. doi: 10.3346/jkms.2011.26.4.561. Epub 2011 Mar 28. PMID 21468265
- [Background] Shim KN, Kim JI, Kim N, Kim SG, Jo YJ, Hong SJ, Shin JE, Kim GH, Park KS, Choi SC, Kwon JG, Kim JH, Kim HJ, Kim JW. The efficacy and safety of irsogladine maleate in nonsteroidal anti-inflammatory drug or aspirin-induced peptic ulcer and gastritis. Korean J Intern Med. 2019 Sep;34(5):1008-1021. doi: 10.3904/kjim.2017.370. Epub 2018 Jun 1. PMID 29847892
- [Background] Julious S. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceut Statist. 2005;4:287-291.
- [Background] Kim HK, Kim JI, Kim JK, Han JY, Park SH, Choi KY, Chung IS. Preventive effects of rebamipide on NSAID-induced gastric mucosal injury and reduction of gastric mucosal blood flow in healthy volunteers. Dig Dis Sci. 2007 Aug;52(8):1776-82. doi: 10.1007/s10620-006-9367-y. Epub 2007 Apr 5. PMID 17410467